CLINICAL TRIAL: NCT05868915
Title: A Phase I/II Clinical Study on the Safety, Tolerability, and Preliminary Efficacy of HV-101 Injection for the Patients With Recurrent or Metastatic Solid Tumors
Brief Title: HV-101 for Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Portfolio prioritization
Sponsor: Hervor Therapeutics (Industry)
Collaborators: Renmin Hospital of Wuhan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CV101
Record Dates: First submitted 2023-05-11; First posted 2023-05-22 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HV-101 (Experimental): Participants with Advanced Solid Tumors
  Interventions:
  Biological: HV-101
  Drug: IL-2
  Drug: Fludarabine Drug: Cyclophosphamide
  Interventions: Biological: HV-101

INTERVENTIONS:
Biological: HV-101 — Biological: HV-101
  HV-101 is autologous tumor-infiltrating lymphocyte cells without genetic modification.
  Drug: IL-2
  Following cell infusion, the patient receives intravenous IL-2.
  Drug: Fludarabine
  Part of the non-myeloablative lymphocyte-depleting preparative regimen.
  Drug: Cyclophosphamide
  Part of the non-myeloablative lymphocyte-depleting preparative regimen.

SUMMARY:
Background:

Tumor-infiltrating lymphocyte (TIL) therapy is a type of adoptive cellular therapy by harvesting infiltrated lymphocytes from tumors, culturing and amplifying them in vitro and then infusing back to treat patients. TIL therapy has shown strong efficacy for the treatment of solid tumors, and has achieved high objective response rates in multiple cancers.

Objective:

To evaluate the safety and efficacy of HV-101 for the treatment of advanced solid tumors.

Eligibility:

Adults aging 18-75 with advanced solid tumors

Design:

1. Patients will undergo screening tests, including imaging procedures, heart and lung tests, and lab tests.
2. Freshly resected patient tumors were dissected by the surgeon.
3. TIL cells were isolated from the patient's tumor tissue in the laboratory, then cultured in vitro, activated and expanded.
4. HV-101 will be re-infused into the patient.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to understand and sign the Informed of Consent Document. Be willing to follow the procedure and protocol of the clinical trial.
2. Age ≥ 18 years and ≤ 75 years.
3. Expected survival time > 3 months.
4. ECOG score 0-1.
5. At least one lesion that could undergo surgery or biopsy to obtain tumor tissue for TIL preparation
6. At least 1 measurable lesion (according to RECIST v1.1).
7. Metastatic or recurrent solid tumors confirmed by histopathology. Refractory to standard treatment evaluated by radiological assessment.
8. Hematology should at least meet the following criteria:

   * Absolute neutrophil count (ANC) ≥ 1.5× 109/L；
   * Platelet (PLT） ≥ 75× 109/L；
   * Hemoglobin (HGB) ≥ 90 g/L.
9. Liver and kidney function are normal:

   * Serum creatinine (Cr) ≤ 1.5 times of upper limit of normal (ULN) or creatine clearance ≥ 60 ml/min;
   * Serum Alanine aminotransferase (ALT) or/and Aspartate aminotransferase (AST) ≤ 2.5 times of ULN;
   * Total bilirubin (TBIL) ≤ 1.5 times of ULN.
10. Blood coagulation function is normal:

    * Prothrombin time (PT) ≤ 1.5 ULN;
    * International Normalized Ratio (INR) ≤ 1.5 ULN;
    * or Activated Partial Thromboplastin Time (APTT) ≤ 1.5 ULN.
11. Women of childbearing potential should be ascetic or take contraception since the signing of ICF to 24 weeks or later after the last administration of drug.

Exclusion Criteria:

1. Under pregnancy or lactation, or positive based on blood pregnancy test.
2. Severe allergic to related ingredients in the clinical trial.
3. Received any other investigational treatment within 28 days before the administration of HV-101.
4. History of other known malignant tumors within the previous 5 years.
5. Primary central nerve system (CNS) cancer, or Participants with CNS metastasis after localized treatment.
6. Participants with any active autoimmune disease, a history of autoimmune disease, or a history or syndrome requiring treatment with systemic steroids or immunosuppressive drugs.
7. Immunodeficiency including HIV positive, acquired or primary immunodeficiency.
8. Participants with ≥ grade 3 thromboembolic events within 6 months or under thrombolysis treatment.
9. Participants with hereditary or acquired hemorrhagic disease.
10. Participants with clinical cardiovascular disease or symptoms
11. Participants with active infection.
12. Participants with active pulmonary tuberculosis infection.
13. Participants with positive hepatitis B surface antigen or positive hepatitis B core antibody or positive hepatitis C virus antibody.
14. Treponema pallidum antibody positive.
15. Participants received major surgery or under severe injury within 28 days before HV-101 infusion.
16. Participants who received live vaccine or attenuated live vaccine 28 days before HV-101 infusion.
17. Participants who have drug addiction history, alcoholism, or drug users.
18. Participants who received cell therapy before enrollment.
19. Participants who have contraindications to the treatment of IL-2 injection.
20. Participants not suitable for the clinical trial evaluated by the investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-08-04 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2026-01-15 (Actual)

PRIMARY OUTCOMES:
Safety of HV-101 | Day 0 - Day 730
  The safety of HV-101 will be assessed based on the totality of dose-limiting toxicity (DLT) and adverse event (AE) data collected during this phase.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Day 0 - Day 730
  To evaluate the proportion of participants who have a confirmed partial response (PR) and complete response (CR) per RECIST v1.1 as assessed by the investigator.
Duration of Response (DOR) | Day 0 - Day 730
  To evaluate the duration from the time that criteria are met for CR or PR per RECIST v1.1 as assessed by the investigator until disease progression or death due to any cause.
Disease Control Rate (DCR) | Day 0 - Day 730
  To evaluate the percentage of participants with a best overall confirmed response of CR or PR at any time plus stable disease (SD) per RECIST v1.1 as assessed by the investigator.
Progression free survival (PFS) | Day 0 - Day 730
  To evaluate the time from the date of HV-101 infusion until disease progression per RECIST v1.1 as assessed by the investigator or death due to any cause.
Overall survival (OS) | Day 0 - Day 730
  To evaluate the time from the date of HV-101 infusion to death due to any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Renmin Hospital of Wuhan University, Wuhan, Hubei, China